CLINICAL TRIAL: NCT04155008
Title: Assessing Quality of Life and the Feasibility of a Nutrition and Pharmacological Algorithm for Oncology Patients With Anorexia
Brief Title: Nutrition and Pharmacological Algorithm for Oncology Patients Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was closed after 4 months due to slow to accrual. Only 1 participant was enrolled.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-10218
Record Dates: First submitted 2019-10-31; First posted 2019-11-07 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Oncologic Complications; Quality of Life; Nutrition Poor; Head and Neck Cancer; Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Malnutrition; Head and Neck Neoplasms; Lung Neoplasms; Pancreatic Neoplasms | interventions — Dexamethasone; Dronabinol; Mirtazapine; Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients with fair to good appetite (Active Comparator): The patients with fair-good appetite (score on CNAQ more than 24) will not receive any pharmacological agents and will receive nutrition intervention alone.
  CNAQ = Council on Nutrition Appetite Questionnaire
  Interventions: Behavioral: Nutrition Intervention
- Patients with poor to fair appetite (Experimental): The patients with poor-fair appetite (score on CNAQ less than 24) will be provided nutrition intervention by the Registered Dietitian and then put into one of three pharmacological groups.
  CNAQ = Council on Nutrition Appetite Questionnaire
  Interventions: Drug: Dexamethasone; Drug: Dronabinol; Drug: Mirtazapine; Behavioral: Nutrition Intervention

INTERVENTIONS:
Drug: Dexamethasone — If the patient's prognosis is extremely poor (less than 12 weeks expected survival, based on discussion with the patient's treating physicians) and there is no additional disease modifying therapy planned, the patient will be prescribed 4mg dexamethasone (which is FDA approved), once daily, to be taken orally in the morning.
  Arms: Patients with poor to fair appetite
Drug: Dronabinol — If the patient has a history of marijuana use or has tried it in the past and had a positive experience with it, then the patient will be prescribed dronabinol (which is FDA approved) 2.5mg, twice daily before meals.
  Other Names: Marinol
  Arms: Patients with poor to fair appetite
Drug: Mirtazapine — If the patient does not have any history of marijuana use, mirtazapine will be prescribed. If the patient is under the age of 70, then the patient would be prescribed 15mg of mirtazapine (which is FDA approved), once daily, to be taken orally at bedtime. For geriatric population (if the patient is over the age of 70), then the patient would be prescribed 7.5mg of mirtazapine, once daily to be taken orally at bedtime.
  Arms: Patients with poor to fair appetite
Behavioral: Nutrition Intervention — Nutrition intervention will be in accordance with the Academy of Nutrition and Dietetics guidelines. The intervention will involve "purposefully planned action(s) designed with the intent of changing a nutrition-related behavior, risk factor, environmental condition, or aspect of health status

SUMMARY:
Loss of appetite is a common symptom of patients with cancer and can cause distress which impacts patients and caregivers. Patients diagnosed with head/neck, lung or pancreatic cancer will be recruited for this study to decrease the suffering and distress associated with eating during cancer treatment and improve the quality of life of patients by implementing an algorithm utilizing nutrition intervention and appetite stimulants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of head/neck, lung, pancreatic cancer, or metastatic cancer from any solid tumor
2. Planned, ongoing, or recently treated patient (within the past 30 days) with chemotherapy, immunotherapy, and/or intravenous targeted biologic therapy
3. No previous use of appetite stimulants
4. All patients must sign study specific informed consent prior to being included in the study
5. No contraindication to appetite stimulants

Exclusion Criteria:

1. Patient <18 years old
2. Contraindication to appetite stimulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Tang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swan WI, Vivanti A, Hakel-Smith NA, Hotson B, Orrevall Y, Trostler N, Beck Howarter K, Papoutsakis C. Nutrition Care Process and Model Update: Toward Realizing People-Centered Care and Outcomes Management. J Acad Nutr Diet. 2017 Dec;117(12):2003-2014. doi: 10.1016/j.jand.2017.07.015. Epub 2017 Oct 5. No abstract available. PMID 28988837
- [Background] Janda M, DiSipio T, Hurst C, Cella D, Newman B. The Queensland Cancer Risk Study: general population norms for the Functional Assessment of Cancer Therapy-General (FACT-G). Psychooncology. 2009 Jun;18(6):606-14. doi: 10.1002/pon.1428. PMID 18942661
- [Background] Doll KM, Kalinowski AK, Snavely AC, Irwin DE, Bensen JT, Bae-Jump VL, Kim KH, Van Le L, Clarke-Pearson DL, Gehrig PA. Obesity is associated with worse quality of life in women with gynecologic malignancies: an opportunity to improve patient-centered outcomes. Cancer. 2015 Feb 1;121(3):395-402. doi: 10.1002/cncr.29061. Epub 2014 Sep 23. PMID 25250951
- [Background] Dapueto JJ, Francolino C, Servente L, Chang CH, Gotta I, Levin R, Abreu Mdel C. Evaluation of the Functional Assessment of Cancer Therapy-General (FACT-G) Spanish Version 4 in South America: classic psychometric and item response theory analyses. Health Qual Life Outcomes. 2003 Aug 20;1:32. doi: 10.1186/1477-7525-1-32. PMID 12969512
- [Background] Sim BY, Lee YW, Kim H, Kim SH. Post-traumatic growth in stomach cancer survivors: Prevalence, correlates and relationship with health-related quality of life. Eur J Oncol Nurs. 2015 Jun;19(3):230-6. doi: 10.1016/j.ejon.2014.10.017. Epub 2014 Dec 18. PMID 25533806
- [Background] Alvarez-Camacho M, Martinez-Michel L, Gonella S, Scrimger RA, Chu KP, Wismer WV. Physical symptom burden of post-treatment head and neck cancer patients influences their characterization of food: Findings of a repertory grid study. Eur J Oncol Nurs. 2016 Jun;22:54-62. doi: 10.1016/j.ejon.2016.03.008. Epub 2016 Apr 7. PMID 27179893
- [Background] Holm T, Maier A, Wicks P, Lang D, Linke P, Munch C, Steinfurth L, Meyer R, Meyer T. Severe loss of appetite in amyotrophic lateral sclerosis patients: online self-assessment study. Interact J Med Res. 2013 Apr 17;2(1):e8. doi: 10.2196/ijmr.2463. PMID 23608722
- [Background] Mattox TW. Cancer Cachexia: Cause, Diagnosis, and Treatment. Nutr Clin Pract. 2017 Oct;32(5):599-606. doi: 10.1177/0884533617722986. Epub 2017 Aug 21. PMID 28825869
- [Background] Cox S, Powell C, Carter B, Hurt C, Mukherjee S, Crosby TD. Role of nutritional status and intervention in oesophageal cancer treated with definitive chemoradiotherapy: outcomes from SCOPE1. Br J Cancer. 2016 Jul 12;115(2):172-7. doi: 10.1038/bjc.2016.129. Epub 2016 Jun 21. PMID 27328311
- [Background] Ravasco P, Monteiro-Grillo I, Marques Vidal P, Camilo ME. Impact of nutrition on outcome: a prospective randomized controlled trial in patients with head and neck cancer undergoing radiotherapy. Head Neck. 2005 Aug;27(8):659-68. doi: 10.1002/hed.20221. PMID 15920748
- [Background] Isenring EA, Capra S, Bauer JD. Nutrition intervention is beneficial in oncology outpatients receiving radiotherapy to the gastrointestinal or head and neck area. Br J Cancer. 2004 Aug 2;91(3):447-52. doi: 10.1038/sj.bjc.6601962. PMID 15226773

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Fair to Good Appetite: The patients with fair-good appetite (score on CNAQ > 24) will not receive any pharmacological agents and will receive nutrition intervention alone.
  Nutrition Intervention: Nutrition intervention will be in accordance with the Academy of Nutrition and Dietetics guidelines. The intervention will involve "purposefully planned action(s) designed with the intent of changing a nutrition-related behavior, risk factor, environmental condition, or aspect of health status
  CNAQ = Council on Nutrition Appetite Questionnaire
- Patients With Poor to Fair Appetite: Patients with poor-fair appetite (score on CNAQ < 24) will be provided nutrition intervention by the Registered Dietitian and then put into one of three pharmacological groups.
  Dexamethasone: If the patient's prognosis is extremely poor (<12 weeks expected survival, based on discussion with the patient's treating physicians) and there is no additional disease modifying therapy planned, the patient will be prescribed 4mg dexamethasone (FDA approved), once daily, to be taken orally in the morning.
  Dronabinol: If the patient has a history of marijuana use or has tried it in the past and had a positive experience with it, then the patient will be prescribed dronabinol (FDA approved) 2.5mg, twice daily before meals.
  Mirtazapine: If the patient does not have any history of marijuana use, mirtazapine will be prescribed. If the patient is under the age of 70, then the patient would be prescribed 15mg of mirtazapine (FDA approved), once daily, to be taken orally at bedtime. For geriatric population (if the patient is over the age of 70), then the patient would be prescribed 7.5mg of mirtazapine, once daily to be taken orally at bedtime.
  Nutrition Intervention: Nutrition intervention will be in accordance with the Academy of Nutrition and Dietetics guidelines. The intervention will involve "purposefully planned action(s) designed with the intent of changing a nutrition-related behavior, risk factor, environmental condition, or aspect of health status
Period: Overall Study
Arm/Group | Patients With Fair to Good Appetite | Patients With Poor to Fair Appetite
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled in this study.
Groups:
- Patients With Fair to Good Appetite: The patients with fair-good appetite (score on CNAQ > 24) will not receive any pharmacological agents and will receive nutrition intervention alone.
  Nutrition Intervention: Nutrition intervention will be in accordance with the Academy of Nutrition and Dietetics guidelines. The intervention will involve "purposefully planned action(s) designed with the intent of changing a nutrition-related behavior, risk factor, environmental condition, or aspect of health status
- Patients With Poor to Fair Appetite: The patients with poor-fair appetite (score on CNAQ < 24) will be provided nutrition intervention by the Registered Dietitian and then put into one of three pharmacological groups.
  Dexamethasone: If the patient's prognosis is extremely poor (<12 weeks expected survival, based on discussion with the patient's treating physicians) and there is no additional disease modifying therapy planned, the patient will be prescribed 4mg dexamethasone (FDA approved), once daily, to be taken orally in the morning.
  Dronabinol: If the patient has a history of marijuana use or has tried it in the past and had a positive experience with it, then the patient will be prescribed dronabinol (FDA approved) 2.5mg, twice daily before meals.
  Mirtazapine: If the patient does not have any history of marijuana use, mirtazapine will be prescribed. If the patient is under the age of 70, then the patient would be prescribed 15mg of mirtazapine (FDA approved), once daily, to be taken orally at bedtime. For geriatric population (if the patient is over the age of 70), then the patient would be prescribed 7.5mg of mirtazapine, once daily to be taken orally at bedtime.
  Nutrition Intervention: Nutrition intervention will be in accordance with the Academy of Nutrition and Dietetics guidelines. The intervention will involve "purposefully planned action(s) designed with the intent of changing a nutrition-related behavior, risk factor, environmental condition, or aspect of health status
- Total: Total of all reporting groups
Arm/Group | Patients With Fair to Good Appetite | Patients With Poor to Fair Appetite | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Assessment
Description: The primary outcome of this study is assessing the impact on quality of life for the oncology patients by using an algorithm for nutrition intervention and appetite stimulants through utilizing Functional Assessment of Cancer Therapy-General Population (FACT-GP).
Time Frame: 3 months
Population: Only 1 patient was enrolled into the study prior to termination. This patient was enrolled into the 'Patients with poor to fair appetite' arm based on their CNAQ score. Data were not collected.
Arm/Group | Patients With Fair to Good Appetite | Patients With Poor to Fair Appetite
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life/Appetite Assessment
Description: The secondary outcome of this study is assessing the impact on quality of life/appetite for the oncology patients by using an algorithm for nutrition intervention and appetite stimulants through utilizing the Council of Nutrition appetite questionnaire.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Patients With Fair to Good Appetite | Patients With Poor to Fair Appetite
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: This was not a therapeutic trial and as such regular review of study conduct, adverse events, and results by a Data and Safety Monitoring Board (DSMB) was not required, and deaths, serious adverse events, and nonserious adverse events were not assessed for planned study participants. As noted only one participant was enrolled into the study.
Arm/Group | Patients With Fair to Good Appetite | Patients With Poor to Fair Appetite
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The primary and secondary outcomes were unable to be assessed as only 1 patient (out of a planned 30) was enrolled into the study. No analyses were therefore conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04155008/Prot_SAP_ICF_000.pdf